CLINICAL TRIAL: NCT01244776
Title: Transplantation of Acellular Corneal Matrix to Treat Corneal Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaanxi Aierfu Activtissue Engineering (Industry)
Collaborators: Shenzhen AiNear Cornea Engineering Company Limited (Unknown); Air Force Military Medical University, China (Other); Engineering Technology Center for Tissue Engineering of Xi'an (Unknown); Beijing Tongren Hospital (Other); West China Hospital (Other); Henan Provincial People's Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Southwest Hospital, China (Other)
Responsible Party: youngbo lu, Shaanxi Aierfu Activtissue Engineering
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEC 01
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Corneal Ulcer
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acellular corneal matrix (Experimental)
  Interventions: Device: acellular corneal matrix

INTERVENTIONS:
Device: acellular corneal matrix — Efficacy of acellular corneal matrix to restore stroma integrity and treat corneal ulcer after lamellar keratoplasty.
  Other Names: ACM

SUMMARY:
This study is to develop a lamellar keratoplasty method for corneal ulcer using acellular corneal matrix (ACM) and to make an analysis among patients for its therapeutic effect.

DETAILED DESCRIPTION:
Infections, chemical injury, and other diseases result in acute or chronic corneal ulcer, which may damage corneal stroma and may lead to permanent corneal scars and blindness. Corneal transplantation is standard method for corneal ulcer, but severe shortage of donor corneas limits its application. Acellular porcine corneal matrix is similar to the native cornea, especially with the biological property and microstructure. Recently, this matrix has been proved to be safe when transplanted to animal subjects and will not be rejected by the recipient. In animal lamellar keratoplasty experiments, acellular corneal matrix showed that they can integrate into the corneal wound bed and help reconstruction of the lamellar integrity of corneal stroma. This study will investigate its healing effect on human corneal ulcer. It will provide a potential corneal substitute for this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 yrs.
* Corneal ulcer.
* Informed consent.

Exclusion Criteria:

* Corneal perforation.
* Other ocular diseases.
* The presence of systemic connective tissue diseases
* Severe allergic constitution
* Pregnancy
* The presence of chronic disease, such as significant cardiovascular illness
* The patients who received clinical experiments for other medicine or medical devices within 3 months prior to the transplantation.
* Any patient that is not suitable for recruitment, in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Rejection evaluation | 30 days following transplantation

SECONDARY OUTCOMES:
Corneal wound healing | 90 days following transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Liuhe Zhou, M.D., Principal Investigator — Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China